CLINICAL TRIAL: NCT04791202
Title: Hypertonic Dextrose Versus Corticosteroid Intra-Articular Injections for the Treatment of Trapeziometacarpal Arthritis: A Prospective Double-blind Randomized Controlled Clinical Trial
Brief Title: Hypertonic Dextrose Versus Corticosteroid Intra-Articular Injections for the Treatment of Trapeziometacarpal Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Collaborators: Kleinert, Kutz and Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20.0174
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pain; Satisfaction, Patient; Functionality
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Glucose; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The clinical assessor is blinded to the baseline evaluations and to the administered treatments. Information about the medications used in the study will be given to the participants, but they will be blinded to their group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dextrose Group (Experimental): Injection for Group A: A 27-gauge needle to be inserted in the 1st CMC joint, at which time 0.5 ml of 15% dextrose mixed with 0.5 ml of 1% lidocaine solution is injected into intra and peri-articular area.
  Interventions: Drug: Dextrose
- Methylprednisolone Acetate Group (Active Comparator): Injection for Group B: A 27-gauge needle to be inserted in the 1st CMC joint, at which time 0.5 ml of 40mg methylprednisolone acetate mixed with 0.5 ml of 1% lidocaine solution is injected into intra and peri-articular area.
  Interventions: Drug: Methylprednisolone Acetate 40 MG/ML

INTERVENTIONS:
Drug: Dextrose — See arm descriptions
  Arms: Dextrose Group
Drug: Methylprednisolone Acetate 40 MG/ML — See arm descriptions
  Arms: Methylprednisolone Acetate Group

SUMMARY:
The evolving reports form recent studies are creating a promise on the potential use of dextrose injections for treating arthritis and replacing current method of treating early osteoarthritis by corticosteroids by giving long standing effect and improving patients' symptoms and function. Over the past 5 years, an increasing number of level I and level II studies have emerged, examining the effect of intra-articular prolotherapy for the treatment of both hip and knee osteoarthritis. On the contrary, there is limited data in small joints, such as the temporomandibular joint.

DETAILED DESCRIPTION:
Carpometacarpal osteoarthritis (OA) is a degenerative condition of the hand that causes pain, stiffness and weakness. It is the second most common site of degenerative disease in the hand after arthritis of the distal interphalangeal joints. The prevalence of symptomatic hand OA in people over 70 years of age has been estimated as 13.4 % for men and 26.2 % for women. OA is more frequent in older age groups, leading to considerable disability with a burden on health services and on the economy. Risk factor for carpometacarpal osteoarthritis of the thumb includes being female, middle age, previous trauma, repetitive use and inflammatory joint disease. Lifetime prevalence of this condition approaches 10%.

Injections are a useful conservative treatment modality prior to considering surgical treatment. Corticosteroid injection is helpful in the treatment of the disease, but some patients gain only short-term benefits. Evolving reports are showing promising results for the application of dextrose as an alternative method for the treatment of Carpometacarpal osteoarthritis, based on their induction for growth factors and inflammatory mediators. For instance, prolotherapy has been used as a treatment of musculoskeletal pain with various etiologies. It has been suggested that prolotherapy induces little inflammation and stimulates endogenous repair especially by prompting release of growth factors. Dextrose is an agent commonly used for prolotherapy.

The evolving reports form recent studies are creating a promise on the potential use of dextrose injections for treating arthritis and replacing current method of treating early OA by corticosteroids by giving long standing effect and improving patients' symptoms and function. Over the past 5 years, an increasing number of level I and level II studies have emerged, examining the effect of intra-articular prolotherapy for the treatment of both hip and knee osteoarthritis. On the contrary, there is limited data in small joints, such as the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria:

* Those patients with diagnosis of carpometacarpal (CMC) osteoarthritis
* Those patients who fit the age limits

Exclusion Criteria:

* Those patients outside of the age limits
* Those patients with systemic rheumatic disease, comorbid hand conditions (such as carpal tunnel syndrome or De Quervain's tenosynovitis), gout, pseudogout
* Those patients with a predisposition to bleeding issues
* Those patients with previous surgery to the affected thumb
* Those patients with previous injection to the involved thumb base within the past 12 months
* Those patients with severe X-ray osteoarthritis of grade IV (Eaton and Littler classification) and no evidence of CMC joint space narrowing on plain radiographs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
post-injection pain | 1 day
  visual analog score for pain (0 for no pain, 10 for worst pain)
post-injection functionality | 1 day
  Q-DASH score for functionality (0 for no disability, 100 for most disability)

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Ozyurekoglu, MD, Principal Investigator — President

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cook GS, Lalonde DH. MOC-PSSM CME article: Management of thumb carpometacarpal joint arthritis. Plast Reconstr Surg. 2008 Jan;121(1 Suppl):1-9. doi: 10.1097/01.prs.0000294708.70340.8c. PMID 18182958
- [Result] Merritt MM, Roddey TS, Costello C, Olson S. Diagnostic value of clinical grind test for carpometacarpal osteoarthritis of the thumb. J Hand Ther. 2010 Jul-Sep;23(3):261-7; quiz 268. doi: 10.1016/j.jht.2010.02.001. Epub 2010 May 10. PMID 20452743
- [Result] van Saase JL, van Romunde LK, Cats A, Vandenbroucke JP, Valkenburg HA. Epidemiology of osteoarthritis: Zoetermeer survey. Comparison of radiological osteoarthritis in a Dutch population with that in 10 other populations. Ann Rheum Dis. 1989 Apr;48(4):271-80. doi: 10.1136/ard.48.4.271. PMID 2712610